CLINICAL TRIAL: NCT00464022
Title: Carbon Dioxide Versus Air Insufflation in Double-Balloon Endoscopy -a Randomised Controlled Multicentre Trial
Brief Title: CO2 Insufflation During Double Balloon Enteroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rikshospitalet University Hospital (Other)
Collaborators: University Hospital Muenster (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2006-3277
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2007-10-17 (Estimated); Status verified 2007-10

CONDITIONS: Pain
Keywords: pain, endoscopy; Pain, endoscopy, randomised trial
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Carbon dioxide

SUMMARY:
Double-balloon enteroscopy (DBE) is a novel endoscopic procedure for visualising the entire small bowel. In any GI endoscopy procedure it is mandatory to insufflate gas into the bowel to secure good visualisation. All endoscopes used for GI endoscopy provide a gas insufflation unit. Currently, air is used for this purpose in more than 90% of centres throughout the world. The use of air, however, is far from ideal to use for insufflation in GI endoscopy. After GI endoscopy, significant amounts of air are usually retained in the bowel segment inspected (5). This air has to pass the GI tract and exit physiologically through the rectum. Thus, abdominal pain and discomfort during and after the examination due to the retention of air has been shown to be very common during and after endoscopic procedures (5-9).

Carbon dioxide gas (CO2), unlike air, is rapidly absorbed from the bowel. Within minutes, several litres of CO2 can be absorbed from the GI tract. The use of CO2 has been shown to result in more comfortable examinations in both colonoscopy and flexible sigmoidoscopy in several randomised trials (6-9). In these studies, CO2 insufflation almost completely reduced procedure-related pain and discomfort.

To our knowledge, no research has been performed investigating the use of CO2 in DBE. DBE is a long-lasting procedure (mean examination time 75 minutes (4)). Large volumes of air are insufflated during the procedure, leading to significant distension of the small bowel during and after the examination.

One of the main technical difficulties in DBE is the formation of small bowel loops and scarp angels during deep intubation of the endoscope. These loops and angels are the major restriction to deep intubation of the endoscope. Loops and scarp angels are more pronounced in air-distended bowel segments.

The aim of the present study is to examine whether CO2 insufflation leads to a reduction of abdominal pain in DBE patients. Furthermore, we want to investigate if CO2 insufflation facilities a deeper intubation of the endoscope and thus a more complete examination of the small bowel mucosa.

The study is designed as a two-centre randomised controlled trial. Randomisation to the two treatment groups (CO2 or air insufflation) is performed on basis of the individual participant.

DETAILED DESCRIPTION:
Background The small bowel has been a large blind spot for gastrointestinal (GI) endoscopy as, until recently, the small bowel was not accessible with conventional endosocopes.

Double-balloon enteroscopy (DBE) is a novel endoscopic procedure for visualising the entire small bowel. The method was first described by Yamamoto et al. and May et al in 2001 and 2003, respectively (1,2). Since then, DBE has spread to a rising number of centres around the world. Both endoscopic diagnosis (e.g. by biopsy) and treatment can be easily performed using DBE. The first larger series, recently published, demonstrate that DBE is feasible in scoping large parts of the small bowel, with total small intubation possible in about 30-40% of cases (3,4).

In any GI endoscopy procedure it is mandatory to insufflate gas into the bowel to secure good visualisation. All endoscopes used for GI endoscopy provide a gas insufflation unit. The gas is pumped on demand into the area examined by the endoscopist via a gas tube incorporated in the endoscope. Currently, air is used for this purpose in more than 90% of centres throughout the world. The use of air, however, is far from ideal to use for insufflation in GI endoscopy. After GI endoscopy, significant amounts of air are usually retained in the bowel segment inspected (5). This air has to pass the GI tract and exit physiologically through the rectum. Thus, abdominal pain and discomfort during and after the examination due to the retention of air has been shown to be very common during and after endoscopic procedures (5-9).

Carbon dioxide gas (CO2), unlike air, is rapidly absorbed from the bowel. Within minutes, several litres of CO2 can be absorbed from the GI tract. The use of CO2 has been shown to result in more comfortable examinations in both colonoscopy and flexible sigmoidoscopy in several randomised trials (6-9). In these studies, CO2 insufflation almost completely reduced procedure-related pain and discomfort.

To our knowledge, no research has been performed investigating the use of CO2 in DBE. DBE is a long-lasting procedure (mean examination time 75 minutes (4)). Large volumes of air are insufflated during the procedure, leading to significant distension of the small bowel during and after the examination.

One of the main technical difficulties in DBE is the formation of small bowel loops and scarp angels during deep intubation of the endoscope. These loops and angels are the major restriction to deep intubation of the endoscope. Loops and scarp angels are more pronounced in air-distended bowel segments.

The aim of the present study is to examine whether CO2 insufflation leads to a reduction of abdominal pain in DBE patients. Furthermore, we want to investigate if CO2 insufflation facilities a deeper intubation of the endoscope and thus a more complete examination of the small bowel mucosa.

Hypothesis

1. The use of CO2 in DBE leads to a reduction in abdominal pain for the patient when compared with the use of air.
2. The use of CO2 in DBE leads to deeper intubation when compared to air insufflation.

Methods Study design The study is designed as a two-centre randomised controlled trial. The participating centres are Rikshospitalet University Hospital, Oslo, Norway and University Hospital Muenster, Germany.

Randomisation to the two treatment groups (CO2 or air insufflation) is performed on basis of the individual participant. Equally large groups are randomised, using block randomisation (blocks of six patients) for each of the participating centres. Randomisation (using SPSS statistical software package) is performed by an independent researcher, who is not part of the DBE team.

Individuals eligible for inclusion are patients referred for DBE at the trial centres who do not fulfil one of the following exclusion criteria:

* Age under 16 years
* Inability to understand information for participation
* Refusal of participation

All eligible individuals are informed about the nature of the study. All individuals provide written informed consent before entering the trial. Patients who do not wish to participate in the present trial are treated according to standard procedures (using air insufflation).

All procedures are performed by experienced endoscopists. Both patients and endoscopists are blinded with regard to type of gas used for any particular patient.

Sedation is performed according to current standards at the centres.

Double-balloon procedure DBE is performed using the DBE endoscope system (Fujinon Inc, Japan), as described in the literature (1-4). The DBE endoscope consist of a 200-cm long video endoscope with an outer diameter of 8.5 mm and a flexible overtube with a length of 145 cm and an outer diameter of 12 mm. Latex balloons are attached to both the endoscope and the overtube. These balloons are inflated and deflated during insertion, as described elsewhere in detail (1,2).

Gas insufflation CO2 is insufflated using Fujinons equipment (or other, to be specified) Air is insufflated using the ordinary air inlet system of the endoscope rack. The air inlet button is hidden from the view of the endoscopist to prevent unblinding (technical details to be specified in cooperation with company).

Evaluation of pain and discomfort A questionnaire is used to classify patient pain during and after the procedure. Visual analogue scales (100-mm) are used to quantify abdominal pain during the examination and at 1, 3, 6, and 24 hours after the procedure, as validated in recent studies (7,8). The questionnaire is given to every participant after the procedure, to be filled in the next day, and mailed back to the respective trial centre using prepaid envelopes.

Evaluation of ERCP examination parameters All procedure parameters of interest (e.g. duration, depth of insertion, use of sedatives) are registered by the endoscopist immediately after the examination using the existing GI lab databases.

Ethics The regional ethics committees of the participating centres will be asked for approval of the study protocol.

Power analysis A 15% reduction in mean pain score on VAS is considered to be clinically important to detect. There are no studies available regarding this outcome in DBE. Therefore, pilot study will be performed with 20 included patients in every group (air/CO2). The results of the pilot study will estimate the standard deviation needed to calculate power and thus size of the study.

Ownership Data are owned by the respective centres. Publication of the study results is planned in a peer-reviewed journal. Michael Bretthauer and Dirk Domagk will co-ordinate study design, data generation and analysis and a first manuscript draft. Michael Bretthauer and Dirk Domagk will be the first authors of the planned publication, the other members of the study groups will be co-authors.

Budget All procedures in the present study are performed in ordinary patients, with ordinary staff and endoscopists. Therefore, no extra costs occur for personal. For the purpose of the present study, however, some technical equipment has to be purchased (to be specified).

Financial funding is needed for meetings of the study group and prepaid envelopes.

References

1. Yamamoto, Sekine Y, Saito Y, et al. Total enteroscopy with a non-surgical steerable double-balloon method. Gatrointest Endosc 2001;53:216-20
2. May A, Nachbar L, Wardak A, et al. Double-balloon enteroscopy: preliminary experience in patients with obscure gastrointestinal bleeding or chronic abdominal pain. Endoscopy 2003;35:985-91
3. May A, Nachbar L, Ell C. Double-balloon enteroscopy (push-and-pull enteroscopy) of the small bowel: feasibility and diagnostic and therapeutic yield in patients with suspected small bowel disease. Gastrointest Endoc 2005;62:62-70
4. Ell C, May A, Nachbar L, et al. Push-and pull enteroscopy in the small bowel using the double-balloon technique: results of a prospective European multicenter study. Endoscopy 2005;37:613-6
5. Hussein AMJ. Carbon dioxide insufflation for more comfortable colonoscopy. Gastrointest Endosc 1984; 30:68-70
6. Stevensen GW et al. Pain following colonoscopy: elimination with carbon dioxide. Gastrointet Endosc 1992;38:564-567
7. Bretthauer M, Thiis-Evensen E, Hoff G, et al. A randomized controlled trial to assess the safety and efficacy of carbon dioxide insufflation in colonoscopy. Gut 2002; 50:604-607
8. Bretthauer M, Hoff G, Thiis-Evensen E, et al. Carbon dioxide insufflation reduces discomfort due to flexible sigmoidoscopy in colorectal cancer screening. Scand J Gastroenterol 2002, 37:1103-8
9. Sumanac K, Zealley I, Fox B , et al. Minimizing postcolonoscopy abdominal pain by using CO2 insufflation: a prospective, randomized, double blind, controlled trial evaluating a new commercially available CO2 delivery system. Gastrointest Endosc 2002;56:190-4

Information and consent Research study: Insuflation of carbon dioxide(CO2) in double balloon enteroscopy

Dear patient

You are hereby kindly invited to participate in a research study while undergoing your planned endoscopic investigation of the small bowel (DBE, double balloon enteroscopy)

During this examination, it is common practice to insufflate gas into the small bowel to provide the examiner with an adequate view. At the vast majority of hospitals around the world, ordinary room air is used for insufflation. However, the insufflated air can produce pain and abdominal discomfort for patients during and in the hours after the examination.

There is some evidence that the use of carbon dioxide gas (CO2) instead of air can reduce abdominal pain after examination. In this study, we would like to find out if this is true.

Study participants will be divided by random into a group that receives CO2 during the DBE examination and one group that receives air.

Both the endoscopist and you as a patient do not know which gas is being used. Only the endoscopy assistant knows the type of gas used during your examination. After the examination, you will receive a short questionnaire about any complaints or discomfort, which we would like to ask you to fill in at home and mail back to the hospital.

If you decide not to participate in the study, your examination will be performed with the use of air insufflation (standard method).

The present study has been approved by the ethics committee. All information will be treated strictly confidential and only for research purposes within this study. Participation is free of charge and not mandatory. You may decline your participation at any time.

Yours sincerely

Dr. med. Michael Bretthauer (tlf:)

Written informed consent I hereby declare my participation in the abovementioned research study. I am aware of that participation is voluntary.

Date Signature

Vedlegg C

Carbon dioxide versus air insufflation in double-balloon endoscopy

"Patient questionnaire (Version 300606), Michael Bretthauer

This questionnaire is to be filled in the day after the procedure and to be mailed back to the GI lab.

Patient ID

1. Was the examination any painful??

   Please score the degree of pain with a vertical dash on the scale below, between No pain (left margin) and very heavy pain (right margin).

   No pain Very heavy pain
2. Did you have any abdominal pain or distension after the examination?

Please score the degree of pain with a vertical dash on the scale below, between No pain (left margin) and very heavy pain (right margin).

No pain Very heavy pain

1 hour after the exam

3 hours after the exam

6 hours after the exam

24 hours after the exam

Please use the back of the questionnaire for any comments

ELIGIBILITY:
Inclusion Criteria:

* Indication for DBE

Exclusion Criteria:

* Age under 16 years
* Inability to understand information for participation
* Refusal of participation

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-11; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Abdominal pain and intubation depth

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bretthauer, Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Domagk D, Bretthauer M, Lenz P, Aabakken L, Ullerich H, Maaser C, Domschke W, Kucharzik T. Carbon dioxide insufflation improves intubation depth in double-balloon enteroscopy: a randomized, controlled, double-blind trial. Endoscopy. 2007 Dec;39(12):1064-7. doi: 10.1055/s-2007-966990. PMID 18072057